CLINICAL TRIAL: NCT00853138
Title: Web-based CBT for Children With Chronic Pain
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Seattle Children's Hospital (Other)
Responsible Party: Principal Investigator, Tonya Palermo, Professor, Anesthesiology and Pain Medicine, Seattle Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R21HD050674 (NIH)
Record Dates: First submitted 2009-02-26; First posted 2009-03-02 (Estimated); Last update posted 2015-05-28 (Estimated); Status verified 2015-05

CONDITIONS: Chronic Pain; Headache; Abdominal Pain
Keywords: cognitive-behavioral therapy; chronic pain; randomized controlled trial; pediatrics
MeSH Terms: conditions — Chronic Pain; Headache; Abdominal Pain | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- CBT (Experimental): Cognitive-behavioral therapy delivered via the internet in eight treatment modules for children (education, stress and negative emotions, deep breathing and relaxation, distraction, cognitive skills, sleep hygiene and lifestyle, staying active, relapse prevention) and eight treatment modules for parents (education, stress and negative emotions, operant strategies I, operant strategies II, modeling, sleep hygiene and lifestyle, communication, relapse prevention).
  Interventions: Behavioral: cognitive-behavioral therapy
- SMC (No Intervention): The standard medical care wait-list control group continued with the treatment recommendations proscribed by their pain care team.

INTERVENTIONS:
Behavioral: cognitive-behavioral therapy — In addition to standard medical care, the children and parents in the family CBT condition will also receive education about chronic pain, pain behaviors and operant strategies as well as training in coping skills using an interactive, engaging format on the Internet.
  The Internet site will consist of three main sections: child treatment modules, parent treatment modules, and diary tracking. All users will complete 8 treatment modules (one per week) over the 8-week treatment period. Each module will require approximately 30-40 minutes to complete. There is separate specific content of the intervention for child users and for parent users.
  Assignments are incorporated into each module for the participant to work on during the treatment week.
  Arms: CBT

SUMMARY:
The purpose of this study is to develop and evaluate the feasibility and effectiveness of a web-based (i.e., internet) treatment approach for providing psychological treatment to reduce pain and improve functioning in children and adolescents with chronic pain.

DETAILED DESCRIPTION:
Chronic pain is an important problem for children and adolescents owing to its high prevalence rate and significant impact on children's mood, daily functioning, and overall quality of life. Effective psychological treatments have been developed to change behaviors and thoughts important in the child's ability to cope with chronic pain. However, the majority of children do not have access to these treatments due to a variety of barriers such as geographical distance from pediatric pain treatment centers.

The purpose of this study is to develop a more accessible method of delivering effective psychological treatment to reduce pain and increase function in children. Children with chronic headache, abdominal, or musculoskeletal pain will be randomized to either receive the web-based treatment right away or to be in a wait-list control condition and receive the treatment 8 weeks later. Both groups of children will continue to receive clinical care through specialty medical clinics. Children's level of pain, their ability to perform, daily functional activities, and overall quality of life will be evaluated before treatment begins, immediately after treatment, and at a 3 month follow up.

ELIGIBILITY:
Inclusion Criteria:

* chronic headache, abdominal, and/or musculoskeletal pain present over the previous 3 months
* interference from pain in at least one area of daily functioning.

Exclusion Criteria:

* serious comorbid chronic condition in the patient (e.g., diabetes, cancer)
* non-English speaking
* previous participation in cognitive-behavioral therapy.

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 48 (Actual)
Dates: Start 2007-05; Primary Completion 2009-03 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
activity limitations | immediately post-treatment, 3 month follow-up

SECONDARY OUTCOMES:
parental response to pain behaviors | immediately post-treatment, 3 month follow-up
depressive symptoms | immediately post-treatment, 3 month follow-up
pain intensity | immediately post-treatment, 3 month follow up

CONTACTS AND LOCATIONS:
Overall Officials: Tonya M Palermo, PhD, Principal Investigator — Seattle Children's Hospital

REFERENCES:
- [Result] Palermo TM, Wilson AC, Peters M, Lewandowski A, Somhegyi H. Randomized controlled trial of an Internet-delivered family cognitive-behavioral therapy intervention for children and adolescents with chronic pain. Pain. 2009 Nov;146(1-2):205-13. doi: 10.1016/j.pain.2009.07.034. Epub 2009 Aug 19. PMID 19695776
- [Result] Law EF, Murphy LK, Palermo TM. Evaluating treatment participation in an internet-based behavioral intervention for pediatric chronic pain. J Pediatr Psychol. 2012 Sep;37(8):893-903. doi: 10.1093/jpepsy/jss057. Epub 2012 Apr 17. PMID 22511033